CLINICAL TRIAL: NCT02175888
Title: The Optimization of Bioavailability From Iron Supplements: Examinations of Different Supplementation Regimens Including Hepcidin Profiles
Brief Title: The Optimization of Bioavailability From Iron Supplements: Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FeSupp_Hep-1
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2015-05

CONDITIONS: Iron Deficiency; Anemia; Iron Deficiency Anemia
Keywords: Iron bio availability; Hepcidin; Iron absorption
MeSH Terms: conditions — Iron Deficiencies; Anemia; Anemia, Iron-Deficiency | interventions — Iron

ARMS (2):
- Oral iron supplement every day for 14 days (Experimental): Daily administration of 60 mg iron in form of ferrous sulphate capsules for 14 consecutive days
  Interventions: Dietary Supplement: Daily administration of 60 mg iron in form of ferrous sulphate capsules for 14 consecutive days
- Oral iron supplement every second day for 28 days (Active Comparator): Administrations of 60 mg iron in form of ferrous sulphate capsules on every second day for 28 days
  Interventions: Dietary Supplement: Administrations of 60 mg iron in form of ferrous sulphate capsules on every second day for 28 days

INTERVENTIONS:
Dietary Supplement: Daily administration of 60 mg iron in form of ferrous sulphate capsules for 14 consecutive days
  Arms: Oral iron supplement every day for 14 days
Dietary Supplement: Administrations of 60 mg iron in form of ferrous sulphate capsules on every second day for 28 days
  Arms: Oral iron supplement every second day for 28 days

SUMMARY:
Iron deficiency (ID) with or without anaemia (IDA) is a major public health problem worldwide, especially in women of reproductive age and young children. Iron supplementation is an effective strategy to prevent and treat ID and IDA. There is a lack of data on iron bioavailability from different supplementation regimens and how to optimize bioavailability in a cost-effective and patient-friendly way. The present study will test whether the fractional and total iron absorption from iron supplements (60 mg) administered daily for 14 days differs from that of iron supplements (60 mg) administered every second day for 28 days. The prevailing serum hepcidin concentration (SHep) is the major determinant of iron absorption and erythrocyte iron utilization. Therefore we will monitor SHep during the whole supplementation period. We hypothesize that the fractional and total iron absorption from the daily administration of 60 mg is lower than that from the administration on every second day due to increased SHep levels when supplements are administered daily.

The study will provide important insights about the optimization of iron bioavailability from different supplementation regimens including the performance of SHep, a key regulator of human iron metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 45 years old,
* Serum ferritin levels </=25 µg/L,
* Normal body Mass Index (18.5-26.5 kg/m2),
* Body weight <80 kg,
* Signed informed consent

Exclusion Criteria:

* Anaemia (Hb < 8.0 g/dL),
* Elevated c-reactive protein or alpha1-glycoprotein concentrations >5.0 mg/L, >1.0 g/L, respectively,
* Any metabolic, gastrointestinal kidney or chronic disease such as diabetes, renal failure, hepatic dysfunction, hepatitis, hypertension, cancer or cardiovascular diseases (according to the participants own statement),
* Continuous/long-term use of medication during the whole studies (except for contraceptives),
* Consumption of mineral and vitamin supplements within 2 weeks prior to 1st supplement administration,
* Blood transfusion, blood donation or significant blood loss (accident, surgery) over the past 4 months,
* Earlier participation in a study using stable iron isotopes,
* Known hypersensitivity or allergy to iron supplements,
* Women who are pregnant or breast feeding,
* Intention to become pregnant during the course of the studies,
* Lack of safe contraception, defined as: Female participants of childbearing potential, not using and not willing to continue using a medically reliable method of contraception for the entire study duration, such as oral, injectable, or implantable contraceptives, or intrauterine contraceptive devices, or who are not using any other method considered sufficiently reliable by the investigator in individual cases.
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the studies, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present studies,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2015-10; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Iron bio-availability from oral iron supplementation (%) | up to 4 weeks
  Iron bioavailability will be assessed with stable isotopic labels. The shift in the isotopic ratio in human whole blood will be measured with Inductively coupled plasma mass spectrometry (ICP-MS).
Serum hepcidin concentrations | 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 17, 19, 21, 23, 25 and 27 days

CONTACTS AND LOCATIONS:
Overall Officials: Diego Moretti, PhD, Principal Investigator — Human Nutrition Laboratory, ETH Zurich
Locations (1):
- Human Nutrition Laboratory, Zurich, Switzerland

REFERENCES:
- [Derived] Lazrak M, El Kari K, Stoffel NU, Elammari L, Al-Jawaldeh A, Loechl CU, Yahyane A, Barkat A, Zimmermann MB, Aguenaou H. Tea Consumption Reduces Iron Bioavailability from NaFeEDTA in Nonanemic Women and Women with Iron Deficiency Anemia: Stable Iron Isotope Studies in Morocco. J Nutr. 2021 Sep 4;151(9):2714-2720. doi: 10.1093/jn/nxab159. PMID 34038558
- [Derived] Stoffel NU, Cercamondi CI, Brittenham G, Zeder C, Geurts-Moespot AJ, Swinkels DW, Moretti D, Zimmermann MB. Iron absorption from oral iron supplements given on consecutive versus alternate days and as single morning doses versus twice-daily split dosing in iron-depleted women: two open-label, randomised controlled trials. Lancet Haematol. 2017 Nov;4(11):e524-e533. doi: 10.1016/S2352-3026(17)30182-5. Epub 2017 Oct 9. PMID 29032957